CLINICAL TRIAL: NCT05968404
Title: A Population-based Study of Pediatric Celiac Disease in South Europe
Brief Title: A Population-based Study of Celiac Disease in South Europe in Children Between 1 to 5 Years of Age
Acronym: HNCEL
Status: Completed | Type: Observational
Sponsor: Hospital Mutua de Terrassa (Other)
Collaborators: Centro de Investigación Biomédica en Red de enfermedades hepáticas y digestivas (CIBERehd) (Unknown); Hospital Sant Joan de Deu (Other); Institut Català d'Oncologia (Other); University of Barcelona (Other); Institut d'Investigació Biomèdica de Bellvitge (Other); Catlab (Unknown)
Responsible Party: Sponsor
Other Study IDs: P13001
Record Dates: First submitted 2023-07-21; First posted 2023-08-01 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-07

CONDITIONS: Celiac Disease
Keywords: Celiac Disease; environmental factors; tolerance to gluten
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Celiac disease (CD) was diagnosed for years almost exclusively in children. This is due to the fact that in adulthood it manifests in a much more attenuated form, while the classic form with severe diarrhea, malnutrition and dehydration is observed almost exclusively in children. Classic studies, carried out prior to the widespread use of serology as a CD diagnostic tool, already showed that there is variability in gluten sensitivity and that in a non-negligible proportion of cases (10%) gluten sensitivity appears to be transient. Subsequent studies, including patients diagnosed by serology or population screening studies, suggest that progression to gluten latency or tolerance may occur in a higher proportion of patients, ranging from 20 to 50% depending on the geographical region.

In the first decade of the 2000s, the researchers group performed a prevalence observational cross-sectional study survey in Catalonia (autonomous region in the northeast of Spain) that accurately reflected the distribution of the reference Catalan population in terms of sex and age. The results showed a drastic and significant drop in the prevalence of CD disease in relation to age, with the prevalence of CD in children being 5 times higher than adults (1:71 vs. 1:357). Strikingly, the reduction in prevalence was especially notable in the first 4 years of life.

Two possibilities were proposed to explain this unexpected finding in a disease that is lifelong: 1) The existence of an environmental effect (cohort effect) acting as a disease trigger in early childhood during the study period (e.g., bacterial or viral infections, vaccines, food policies related to gluten introduction, use of antibiotics, etc.). 2) The appearance of age-related tolerance to gluten in a proportion of cases. Interestingly, it has been suggested that immunological tolerance might be more frequent in children diagnosed with CD before the age of two.

The aims of the present epidemiological study are: 1) to determine the prevalence of CD in Catalonia in children under 5 years of age and compare it with the results obtained in the previous 2004-2007 study; 2) to investigate the potential effect of environmental factors on disease prevalence; and 3) to evaluate longitudinally the appearance of tolerance to gluten in the CD cases detected. Therefore, this study has been designed using exactly the same CD screening methodology and reproducing the reference population in the same geographical area as the previous 2004-2007 study.

ELIGIBILITY:
Exclusion Criteria:

* Heart failure or unstable cardiopathy
* COPD or respiratory insufficiency
* Coagulopathy
* Hepatic cirrhosis
* Kidney failure
* Active neoplasm
* Gluten-free diet without CD diagnosis

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Pediatric patients from ambulatory minor surgery departments (= general population sample). Regarding age and sex, inclusion is done reproducing the reference population of the area.
Sampling Method: Probability Sample
Enrollment: 3659 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
CD prevalence | at inclusion
  CD cases detection via tissue transglutaminase IgA antibodies (tTGA)(serological CD marker) in blood serum

REFERENCES:
- [Background] Vivas S, Ruiz de Morales JM, Fernandez M, Hernando M, Herrero B, Casqueiro J, Gutierrez S. Age-related clinical, serological, and histopathological features of celiac disease. Am J Gastroenterol. 2008 Sep;103(9):2360-5; quiz 2366. doi: 10.1111/j.1572-0241.2008.01977.x. Epub 2008 Aug 12. PMID 18702652
- [Background] Ansaldi N, Tavassoli K, Faussone D, Forni M, Oderda G. [Clinico-histological behavior of celiac patients after gluten load following the definitive diagnosis]. Pediatr Med Chir. 1988 Jan-Feb;10(1):3-6. Italian. PMID 3375125
- [Background] Matysiak-Budnik T, Malamut G, de Serre NP, Grosdidier E, Seguier S, Brousse N, Caillat-Zucman S, Cerf-Bensussan N, Schmitz J, Cellier C. Long-term follow-up of 61 coeliac patients diagnosed in childhood: evolution toward latency is possible on a normal diet. Gut. 2007 Oct;56(10):1379-86. doi: 10.1136/gut.2006.100511. Epub 2007 Feb 15. PMID 17303598
- [Background] Marine M, Farre C, Alsina M, Vilar P, Cortijo M, Salas A, Fernandez-Banares F, Rosinach M, Santaolalla R, Loras C, Marques T, Cusi V, Hernandez MI, Carrasco A, Ribes J, Viver JM, Esteve M. The prevalence of coeliac disease is significantly higher in children compared with adults. Aliment Pharmacol Ther. 2011 Feb;33(4):477-86. doi: 10.1111/j.1365-2036.2010.04543.x. Epub 2010 Dec 19. PMID 21166832